CLINICAL TRIAL: NCT03035292
Title: Proof of Concept Trial of a Novel Imaging System to Assess and Document Choroidal Reflectance in Children for the Detection of Cataract and Media Opacities.
Brief Title: Infrared Choroidal Reflectance Camera for the Detection of Childhood Cataract
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Louise Allen, Consultant Paediatric Ophthalmologist, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 159569; REC17/EE/0010 (Other: IRAS)
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-01

CONDITIONS: Childhood Cataract

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children attending eye clinic: Children 1 month to 5 years of age attending paediatric ophthalmology clinic with and without cataracts. Children who had previously had intra-ocular surgery were excluded.
  One eye of each child was assessed by an inexperienced screener (medical student) by red-reflex assessment using direct ophthalmoscope and infrared-reflex using a new device (CatCam). CatCam is a modified smart phone camera which images the reflection of co-axial infrared light from the ocular fundus. A cataract appears as a black silhouette on the white infrared-reflex imaged by the camera.
  Sensitivity and specificity for red-reflex and infrared-reflex assessment compared to gold standard dilated ophthalmic examination by a specialised were compared.
  Interventions: Diagnostic Test: Red-reflex assessment; Diagnostic Test: Infrared-reflex assessment

INTERVENTIONS:
Diagnostic Test: Red-reflex assessment — The red reflex was examined in the standard manner using direct ophthalmoscope by medical student examiner
Diagnostic Test: Infrared-reflex assessment — The infrared reflex was examined using a modified smart phone camera by a medical student examiner

SUMMARY:
Sensitivity and specificity of current screening methods for childhood cataracts is poor. This results in delayed diagnosis and management which can decrease the visual prognosis following cataract surgery. It also results in many false positives with resultant unnecessary healthcare costs in specialist paediatric ophthalmology services. This study compares the accuracy of cataract screening using infrared light compared to white light in a population of children attending eye clinic.

DETAILED DESCRIPTION:
All babies born in the United Kingdom (UK) undergo eye screening to enable the early diagnosis and management of childhood cataract, a treatable but potentially blinding condition affecting 1 in 2000 newborns. The current technique involves the assessment of the "red-reflex" - the orange/red glow in the pupil seen during ophthalmoscopy (or flash photography) due to reflectance of light from the back of the eye. In reality, testing can be technically difficult because the pupil constricts to light during the examination and, particularly in babies of Asian and Afro-Caribbean ancestry, the red-reflex can be dim due to the effect of ocular pigmentation. As a result less than 50% of congenital cataracts are currently identified up by screening. Early visual experience is required for good visual development and a delay in the surgical management of cataracts results in sub-optimal visual development and visual impairment.

There are theoretical advantages to using Infrared (IR) light rather than white light to assess choroidal reflectance, including avoidance of pupil constriction. The study aims to determine if the assessment of the IR-reflex, using a prototype device, rather than the red-reflex, using a direct ophthalmoscope, improves screening accuracy in the detection of ocular media opacities in a pathology enriched childhood cohort.

Eligible children attending an eye clinic will be screened for cataract by a medical student (masked to the pathology) using the existing standard direct ophthalmoscope technique for red-reflex assessment and IR-reflex assessment using the prototype imaging device. A gold standard examination by an ophthalmologist will follow the screening examinations. Sensitivity and specificity of each screening technique will be calculated and compared.

ELIGIBILITY:
Inclusion Criteria:

* All children between 1 month and 5 years of age attending paediatric ophthalmology clinic

Exclusion Criteria:

* Parents / carers with poor conversant English

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and children from 1 month to 5 years of age attending a specialist paediatric ophthalmology clinic with or without known cataracts.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise E Allen, MD, Principal Investigator — Cambridge University Hospitals NHS Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahi JS, Dezateux C. National cross sectional study of detection of congenital and infantile cataract in the United Kingdom: role of childhood screening and surveillance. The British Congenital Cataract Interest Group. BMJ. 1999 Feb 6;318(7180):362-5. doi: 10.1136/bmj.318.7180.362. PMID 9933197
- [Background] Mndeme FG, Mmbaga BT, Kim MJ, Sinke L, Allen L, Mgaya E, Bastawrous A, MacLeod D, Burton MJ, Gilbert C, Bowman R. Red reflex examination in reproductive and child health clinics for early detection of paediatric cataract and ocular media disorders: cross-sectional diagnostic accuracy and feasibility studies from Kilimanjaro, Tanzania. Eye (Lond). 2021 May;35(5):1347-1353. doi: 10.1038/s41433-020-1019-5. Epub 2020 Jun 16. PMID 32546747
- [Result] Duret A, Humphries R, Ramanujam S, Te Water Naude A, Reid C, Allen LE. The infrared reflex: a potential new method for congenital cataract screening. Eye (Lond). 2019 Dec;33(12):1865-1870. doi: 10.1038/s41433-019-0509-9. Epub 2019 Jul 2. PMID 31267092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Diagnostic accuracy comparison trial: children from 1 month to 5 years of age (with no previous history of ophthalmic surgery) attending a specialist paediatric out-patient clinic were enrolled into the study over a 3 month period.
Units Other Than Participants: Eyes
Groups:
- Children Recruited to Diagnostic Comparison Study: Right eyes of children recruited to the study who underwent the following sequential examinations at the time of their clinic appointment: 1) red-reflex assessment by a medical student using direct ophthalmoscope 2) infrared-reflex assessment by the same medical student using the choroidal reflectance imaging device and 3) gold standard ophthalmic examination.
Period: Overall Study
Arm/Group | Children Recruited to Diagnostic Comparison Study
Started | 110; 110 Eyes
Completed | 110; 110 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: Children having red-reflex, infrared-reflex and gold standard examination. Data for the right eye only was analysed.
Units Other Than Participants: Eyes
Groups:
- Children Recruited to Diagnostic Comparison Study: The data from right eyes of 110 children recruited to diagnostic accuracy comparison trial from clinic. These patients had initial red-reflex assessment (Intervention 1) and then infrared-reflex assessment (intervention 2) performed by a medical student prior to gold standard examination by a paediatric ophthalmologist
Arm/Group | Children Recruited to Diagnostic Comparison Study
Number analyzed (Participants) | 110
Number analyzed (Eyes) | 110
Age, Continuous [Median (Standard Deviation); unit: years] | 4 (3.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ethnicity: white | 89
  ethnicity: black, asian, minority ethnic | 21
Evaluator assessment of reflex [Count of Participants; unit: Participants] | 110

OUTCOME MEASURES:

1. Primary Outcome: Results of Red-reflex and Infrared-reflex Tests Compared to Gold Standard
Description: True positives: the number of eyes with cataract correctly identified True negatives: the number of eyes without cataract correctly identified False positives: the number of eyes without cataracts incorrectly identified as having cataract False negatives positives: the number of eyes with cataract incorrectly identified as not having cataract
Time Frame: 1 day
Population: 110 children were eligible for the study, each had their right eye assessed by a medical student using 1) red-reflex assessment 2) Infrared-reflex assessment. Findings were compared to a gold standard examination by an ophthalmologist.
Measure: Number; unit: eyes
Groups:
- Eyes Tested in the Diagnostic Comparison Study: Eyes of children having red-reflex and infrared reflex tests
Arm/Group | Eyes Tested in the Diagnostic Comparison Study
Number analyzed (Participants) | 110
eyes
  Red-reflex test true positive | 17
  Red-reflex test true negative | 54
  Red-reflex test false positive | 32
  Red-reflex test false negative | 7
  Infrared-reflex test true positive | 24
  Infrared-reflex test true negative | 86
  Infrared-reflex test false positive | 0
  Infrared-reflex test false negative | 0

2. Primary Outcome: Sensitivity and Specificity of Red-reflex and Infrared-reflex Testing
Description: Sensitivity (percentage of eyes with cataract correctly identified) and specificity (percentage of eyes without cataract correctly identified) of red-reflex and infrared-reflex testing in percentage terms with 95% Confidence Intervals. Sensitivity and specificity are recorded as a percentage, with 100% indicating best accuracy.
Time Frame: 1 day
Population: 110 eyes (of 110 children) recruited to the study
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Eyes Tested in the Diagnostic Comparison Study: Results of red-reflex, infra-red reflex findings compared to gold standard
Arm/Group | Eyes Tested in the Diagnostic Comparison Study
Number analyzed (Participants) | 110
Number analyzed (Eyes) | 110
percentage of eyes
  Sensitivity of red-reflex | 71 [58 to 89]
  Sensitivity of infrared-reflex | 100 [83 to 100]
  Specificity of red-reflex | 63 [53 to 73]
  Specificity of infrared-reflex | 100 [95 to 100]
Statistical Analysis 1: Comparison: Eyes Tested in the Diagnostic Comparison Study; Sample size was based on a cataract prevalence of 20% in the enriched population and a predicted difference of 15% sensitivity and specificity between tests; Test type: Superiority; p < 0.05, McNemar — This value of <0.05 is the calculated p value where the a priori threshold for statistical significance is considered to be p=0.05

3. Secondary Outcome: Results of Red-reflex and Infrared-reflex Tests Compared to Gold Standard Stratified by Ethnicity
Description: True positives: the number of eyes with cataract correctly identified in caucasian children's eyes and in BAME children's eyes. True negatives: the number of eyes without cataract correctly identified in caucasian children's eyes and in BAME children's eyes. False positives: the number of eyes without cataract incorrectly identified as having cataract in caucasian children's eyes and in BAME children's eyes. False negatives: the number of eyes with cataract incorrectly identified as not having cataract in caucasian children's eyes and in BAME children's eyes.
Time Frame: 1 day
Population: of 110 eligible children, 89 (81%) were caucasian, 21(19%) were of Black, Asian or minority ethnicity (BAME)
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Eyes Tested in the Diagnostic Comparison Study: Eyes of children undergoing red-reflex and infrared-reflex assessment
Arm/Group | Eyes Tested in the Diagnostic Comparison Study
Number analyzed (Participants) | 110
Number analyzed (Eyes) | 110
Eyes
  Red-reflex true positives in BAME children's eyes | 2
  Red-reflex true negatives in BAME children's eyes | 5
  Red-reflex false positives in BAME children's eyes | 14
  Red-reflex false negatives in BAME children's eyes | 0
  Red-reflex true positives in white children's eyes | 15
  Red-reflex true negatives in white children's eyes | 49
  Red-reflex false positives in white children's eyes | 18
  Red-reflex false negatives in white children's eyes | 7
  Infrared-reflex true positives in BAME children's eyes | 2
  Infrared-reflex true negatives in BAME children's eyes | 19
  Infrared-reflex false positives in BAME children's eyes | 0
  Infrared-reflex false negatives in BAME childrens' eyes | 0
  Infrared-reflex true postives in white children's eyes | 22
  Infrared-reflex true negatives in white children's eyes | 67
  Infrared-reflex false positives in white children's eyes | 0
  Infrared-reflex false negatives in white children's eyes | 0

4. Secondary Outcome: Sensitivity and Specificity of Red-reflex and Infrared-reflex Testing Stratified by Ethnicity
Description: as for outcome 2
Time Frame: 1 day
Population: 89 (81%) were the eyes of caucasian children, 21(19%) were the eyes of Black, Asian or minority ethnicity (BAME) children
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Eyes Tested in the Diagnostic Comparison Study: 110 right eyes of 110 children of diverse ethnicity tested with the two fundus reflex techniques. Eyes first underwent red-reflex assessment (Intervention 1) and then infrared-reflex assessment (intervention 2) performed by a medical student prior to gold standard examination by a paediatric ophthalmologist
Arm/Group | Eyes Tested in the Diagnostic Comparison Study
Number analyzed (Participants) | 110
Number analyzed (Eyes) | 110
percentage of eyes
  Sensitivity of red-reflex in caucasian eyes | 69 [49 to 88]
  Sensitivity of red-reflex in BAME eyes | 100 [20 to 100]
  Specificity of red-reflex in caucasian eyes | 72 [61 to 82]
  Specificity of red-reflex in BAME eyes | 32 [11 to 53]
Statistical Analysis 1: Comparison: Eyes Tested in the Diagnostic Comparison Study; Evidence of superiority of intervention 2 over intervention 1 requires a significant difference in specificity of the intervention 1 and 2 between ethnicity groups; Test type: Superiority; p < 0.05, Fisher Exact — The calculated p value was <0.05. A priori threshold for statistical significance is p=0.05

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Children Recruited to Diagnostic Comparison Study: 110 children recruited to diagnostic accuracy comparison trial from clinic. These patients had initial red-reflex and infra-red reflex assessment using an imaging device performed by a medical student prior to gold standard examination by a paediatric ophthalmologist
Arm/Group | Children Recruited to Diagnostic Comparison Study
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT03035292/Prot_SAP_000.pdf